CLINICAL TRIAL: NCT06194591
Title: Low-intensity Extracorporeal Shockwave Therapy With the Nephrospec TM Device for the Treatment of Hypertension in Patients Diagnosed With Chronic Kidney Disease (CKD) : a Randomized, Double-blind Sham-controlled Monocentric Trial
Brief Title: Nephrospec Switzerland
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Menno Pruijm (Other)
Responsible Party: Sponsor-Investigator, Menno Pruijm, Pr., Centre Hospitalier Universitaire Vaudois
Organization: Centre Hospitalier Universitaire Vaudois (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023-D0075
Record Dates: First submitted 2023-12-15; First posted 2024-01-08 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Chronic Kidney Diseases; Hypertension
Keywords: CKD; Chronic Kidney Disease; Hypertension; Li-ESWT; Low-Intensity Extracorporeal Shock Wave Therapy
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension

STUDY DESIGN:
Intervention Model Description: The medical device used to administer Low-intensity extracorporeal shockwave therapy (Li-ESWT) is the NephrospecTM device from Curespec (manufacutred by Medispec). This device is CE-marked, has been used in previous studies, and will be used according to its instructions of use.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A sham device is used. The sham device is visually identical to the NephrospecTM device but disposes of a metal bar that prevents the shockwaves to be transmitted to the patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Stage A - Active treatment (Active Comparator): The medical device NephrospecTM is used to administer 6 treatments of Low-intensity extracorporeal shockwave therapy (Li-ESWT) to the kidneys during 3 weeks.
  Interventions: Device: NephrospecTM, low-intensity extracorporal shockwave therapy device
- Stage A - Sham treatment (Sham Comparator): The sham group will undergo the same treatment schedule, but with an applicator with an internal barrier to prevent shockwaves to pass through to the patient.
  Interventions: Device: Sham-Device
- Stage B - Open label active treatment (Active Comparator): Patients that were in the placebo group of stage A and do not exhibit a significant improvement in one of the main parameters will be eligible to enter stage B where they are treated with the active device in an open-label fashion.
  Interventions: Device: NephrospecTM, low-intensity extracorporal shockwave therapy device

INTERVENTIONS:
Device: NephrospecTM, low-intensity extracorporal shockwave therapy device — Patients will receive 6 Li-ESWT treatments with the NephrospecTM device over three consecutive weeks, with a minimal recess of 24 hours between treatments and a maximum of 3 sessions per week.
  Three hundred shockwaves will be applied by the PI or co-PI to each one of 8 pre-selected regions of each kidney, under ultrasound control, with the patient in the prone position. No local anaesthesia is needed. Total treatment time of one session is 30 minutes. The participant will remain under supervision for another 30 minutes and will be discharged hereafter.
  Arms: Stage A - Active treatment; Stage B - Open label active treatment
Device: Sham-Device — The sham device is the NephrospecTM applicator with an internal barrier to prevent shockwaves to pass through to the patient.
  Arms: Stage A - Sham treatment

SUMMARY:
This is a randomized, double-blind sham-controlled monocentric trial. 30 patients that are diagnosed with hypertension and with moderate to severe chronic kidney disease are included in this trial. 20 of them are randomized into the active treatment arm, 10 into the sham arm. Low-intensity extracorporal shock wave (Li-ESWT) sessions (arm1) or sham sessions (arm2), will be administered with a dedicated probe within three consecutive weeks to the kidneys of patients.The study will add data to the effects of the shock wave treatment on blood pressure and will assess whether this treatment improves renal function, perfusion and oxygenation. The study includes a third arm (arm3) in which treatment sessions are administered to patients that were in the placebo group in the first phase of the study (arm2).

DETAILED DESCRIPTION:
This is a randomized, double-blind sham-controlled monocentric trial. Adult patients that are diagnosed with hypertension (systolic blood pressure 135 - 180 mmHg), currently on stable (over 60 days) medical therapy and with moderate to severe chronic kidney disease (eGFR 20-70 mL/min/1.73m2) or with eGFR between 60-90 ml/min/1.73m 2 and albuminuria ≥30 mg/mmol in spot urine or ≥300 mg/day in 24h urine collection who are currently on stable (at least 60 days) medical therapy are included in this trial.

20 patients are randomized into the active treatment arm with the investigational medical device, 10 patients into the sham arm. Low-intensity extracorporal shock wave (Li-ESWT) sessions (arm1) with a dedicated probe (Nephrospec device) or sham sessions (arm2), within three consecutive weeks, will be applied to the kidneys of patients. Patients will be followed-up for 48 weeks after the treatment.The study includes a third arm (arm3) in which treatment sessions are administered to patients that were in the placebo group in the first phase of the study and for whom their condition did not improve (arm 2).

Low-intensity extracorporeal shockwave therapy (Li-ESWT) is based on the classic technique of lithotripsy for the extracorporeal treatment of kidney stones but applied at much lower intensity (~10%). Previous histological studies in animals have shown that Li-ESWT has favourable effects on kidney perfusion and oxygenation. In human studies that included patients with diabetic nephropathy, six to twelve sessions of Li-ESWT lead to long-term reduction of blood pressure and stabilization of renal function (eGFR). The medical device Nephrospec TM is CE-mark and used in the ambulatory setting to lower BP in patients with CKD. The device will be used according to the instructions and indications mentioned in the operator manual.

The primary outcome of this trial is the change in systolic 24-hour ambulatory blood pressure (ABPM) from baseline to 12 weeks post treatment. Further important secondary ouctomes are automatic office blood pressure (AOBP), the change in number or dose of blood pressure medications, the change in eGFR and the change in albumine/creatinine ratio (ACR). Furthermore, the study will assess whether the treatment improves renal function, Contrast enhanced ultrasound (CEUS)-assessed perfusion index, as well as renal oxygenation and fibrosis (ADC) assessed by MRI.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years to 82 years.
* Patient is diagnosed with Hypertension, i.e. home,office and/or 24h systolic blood pressure ≥135 mmHg (as per ISH guidelines, 2020), currently on stable (over 60 days) medical therapy as prescribed by a physician, of none, one, or more antihypertensive medication classes. Patients will be considered stable if no relevant medication change for over 60 days or for 30 days if there were no previous changes 90 days before the current change.
* Patients diagnosed with moderate to severe chronic renal failure (eGFR 20-70 mL/min/1.73m2) who are currently on stable medical therapy as prescribed by a physician.
* Patients with eGFR between 60-90 ml/min/1.73m2 and albuminuria >=30mg/mmol in spot urine or >=300mg/day in 24h urine collection
* Patient is able and willing to comply with the required follow-up schedule.
* Patient is capable of giving an informed consent.

Exclusion Criteria:

* Hypertension: Individual's systolic BP is over 180mmHg when receiving stable medical medication regimen as prescribed by a physician, of none, one, or more antihypertensive medication classes at maximally tolerated dose. Hypertension secondary to an identifiable and treatable cause, other than Renal artery stenosis or CKD, or is prescribed a medication that may raise BP.
* History of previous renal artery stent. Stent or other intervention involving renal arteries including but not limited to renal denervation procedures.
* Kidney conditions non compatible with the study: Patient has an eGFR <20 ml/min/1.73m², is on Dialysis or has had a kidney transplant performed. Active pyelonephritis. History of or current kidney stones. Patients with polycystic kidney disease or a known complicated renal cyst (Bosniak III or higher).
* Symptomatic patients (Macrohematuria) with a decrease of over 2 grams in Hb.
* Hemoglobin (Hb) ≤ 9 grams per deciliter (blood).
* Coagulation issues: Bleeding tendency resulting from hematologic disease. Subjects having INR > 2.5 and PT, PTT and platelet count which deviates from the clinical laboratory normal reference range.
* Diseases non compatible with the study: Recent (less than 6 months) history of myocardial infarction, PCI, stroke or hospitalization for HFrEF (heart failure with reduced ejection fraction). Individual has type 1 diabetes mellitus or poorly controlled type 2 diabetes mellitus (HbA1c > 10%).
* Active Cancer - primary tumor or metastatic, such as liver, renal, testicular, abdominal tumor or local tumor at treatment area..
* Treatment non compatible with the study: Patients that have been treated with immunosuppression in the last 3 months. Individual requires chronic oxygen support or mechanical ventilation other than nocturnal respiratory support for sleep apnea. No change in dosing of RAS inhibitors in the month prior to the procedure is required.
* Technical impossibility to participate: Local infection of the skin at the area to be in contact with the applicator.
* Known allergy to Sonovue® contrast product (hypersensibility to sulfur hexyfluoride or another component).
* No other contraindication to SonoVue, ie. patients with right-to-left shunts, severe pulmonary hypertension (pulmonary arterial pressure > 90 mm Hg), uncontrolled systemic hypertension and in adult patients with respiratory distress syndrome (ARDS).
* Contraindication to undergo MR-imaging such as the presence of a pacemaker or other implanted metallic device or severe claustrophobia.
* Inability to follow the procedures of the investigation, e.g. due to language problems, psychological disorders, dementia, etc. of the subject/ Unable to obtain consent
* Known or suspected non-compliance, drug or alcohol abuse
* Individual works night shifts.
* Individual is pregnant, breast feeding or planning to become pregnant.
* Individual does not want to be informed in case of accidental finding related to individual's health discovered during imaging or other study-related exams.
* Participation in another investigation with an investigational drug or another MD within the 30 days preceding and during the present investigation,
* Previous enrolment into the current investigation,
* Enrolment of the PI, his/her family members, employees, and other dependent persons

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Systolic 24-hour ambulatory blood pressure (ABPM) | Baseline to 12-weeks (-1/+3weeks) Follow-up post last treatment.
  Assess the Systolic 24-hour ambulatory blood pressure depending on the particpant's arm affiliation

SECONDARY OUTCOMES:
attended Automatic Office Blood Pressure | baseline to 4 weeks (+3 weeks), 24 weeks (±3 weeks) and 48 weeks (±3 weeks) post last treatment
  Assess the attended Automatic Office Blood Pressure depending on the particpant's arm
unattended Automatic Office Blood Pressure | from baseline to 4 weeks (+3 weeks), 24 weeks (±3 weeks) and 48 weeks (±3 weeks) post last treatment
  Assess the unattended Automatic Office Blood Pressure depending on the particpant's arm
Number, dose or number of medications to maintain blood pressure control | baseline to 24 weeks (±3 weeks), and 48 weeks (±3 weeks) post last treatment
  Assess the number, dose or number of medications to maintain blood pressure control depending on the particpant's arm
Serum creatinine levels / eGFR - calculated by CKD - EPI | baseline to 4 weeks (+3 weeks), 12 weeks (-1/+3 weeks), 24 weeks (±3 weeks), and 48 weeks (±3 weeks) post last treatment.
  Assess the serum creatinine levels / eGFR (calculated by CKD - EPI) depending on the particpant's arm
Albumin/creatinine ratio (ACR) | baseline to 4 weeks (+3 weeks), 12 weeks (-1/+3 weeks), 24 weeks (±3 weeks), and 48 weeks (±3 weeks) post last treatment.
  Assess the albumin/creatinine ratio (ACR) depending on the particpant's arm
CEUS-assessed Perfusion Index (PI) | baseline to 12 weeks (±3 weeks)
  Assess the CEUS-assessed Perfusion Index (PI) depending on the particpant's arm
MRI-assessed oxygenation (R2*), fibrosis (ADC) and Phase-contrast | baseline to 12 weeks (±3 weeks)
  Assess the MRI-assessed oxygenation (R2*), fibrosis (ADC) and Phase-contrast depending on the particpant's arm
Plasma renin activity | baseline to 12 weeks (±3 weeks)
  Assess the plasma renin activity depending on the particpant's arm
Plasma aldosterone levels | baseline to 12 weeks (±3 weeks)
  Assess the plasma aldosterone levels depending on the particpant's arm
Cystatin C levels | baseline to 12 weeks (±3 weeks)
  Assess the cystatin C levels depending on the particpant's arm

CONTACTS AND LOCATIONS:
Overall Officials: Menno Pruijm, Dr, Principal Investigator — CHUV
Locations (1):
- Department of Nephrology, Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided